CLINICAL TRIAL: NCT02393326
Title: Biodentine Partial Pulpotomy of Pulpally Exposed Primary Molars
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: technical and funding issues
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Avia Fux, pediatric dentist, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0644-14-HMO-CTIL
Record Dates: First submitted 2015-03-09; First posted 2015-03-19 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Pulpotomy; Tooth, Deciduous
MeSH Terms: interventions — tricalcium silicate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partial pulpotomy with biodentine (Experimental): Biodentine is gently applied to the pulp stumps
  Interventions: Procedure: partial pulpotomy with biodentine
- Formocresol pulpotomy (Other): A cotton pellet moistened with formocresol (1: 5 Buckley's solution) is placed on the amputated pulp for 5 min.
  Interventions: Procedure: Formocresol pulpotomy

INTERVENTIONS:
Procedure: partial pulpotomy with biodentine — After caries removal resulted in a pulp exposure, the pulp at the exposed area is amputated to a depth of 2 mm. The wound surface is irrigated and dried. After homeostasis is obtained, biodentine is gently applied to the wound surface, and then covered with reinforced zinc oxide-eugenol
  Arms: Partial pulpotomy with biodentine
Procedure: Formocresol pulpotomy — Following removal of the coronal pulp and achievement of homeostasis, a cotton pellet moistened with formocresol (1: 5 Buckley's solution) is placed on the amputated pulp for 5 min. The pulp stumps is then covered by IRM.
  Arms: Formocresol pulpotomy

SUMMARY:
Objective: To compare success rates of biodentine partial pulpotomy versus formocresol pulpotomy treatment of pulpally exposed lower primary molars.

After caries removal resulted in a pulp exposure, the pulp at the exposed area is amputated to a depth of 2 mm. The wound surface is irrigated and dried. After homeostasis is obtained, an assistant drew lots to randomly allocate the case to either the biodentine partial pulpotomy (PP) or the formocresol pulpotomy (FP) group.

The follow-up for clinical and radiographic evaluation will be carried out at 6-month intervals.

DETAILED DESCRIPTION:
* Prospective
* Study population: 100 patients.
* Study group: This study sample comprises mandibular primary molars from boys and girls aged between 3 and 7 years. The children have no systemic diseases according to the medical history supplied by the parents or guardians. The mandibular primary molars in this study are selected according to the following clinical and radiographic criteria. The clinical criteria: the presence of a deep carious lesion, sufficient tooth structure for restoration with a stainless steel crown, no history of spontaneous pain, tenderness to percussion or abnormal mobility, abscess, fistula, or swelling of the gingiva, and with cessation of bleeding after a 2 mm depth of the pulp at the area of the exposure was amputated. The radiographic criteria: a deep carious lesion in close proximity to the pulp without furcation or radicular pathology, obliteration of the pulp and root canal, or internal or external root resorption. Physiologic root resorption, while included in the criteria, could not be more than one-third of the root length.
* Clinical technique: All teeth will be treated under local anaesthesia with rubber dam isolation. After caries removal resulted in a pulp exposure, the pulp at the exposed area is amputated to a depth of 2 mm using a water-cooled high-speed handpiece with a #330 high-speed bur. The wound surface is irrigated with sterile saline solution and dried with cotton pellets to avoid clot formation. After homeostasis is obtained, an assistant drew lots to randomly allocate the case to either the PP or the FP treatment group. The child will not know which treatment is assigned to each tooth. For the PP group, biodentine is gently applied to the wound surface, and then covered with reinforced zinc oxide-eugenol (IRM_; Dentsply). For the FP group, coronal access is obtained using high-speed handpiece with a #330 high-speed bur with water spray to further expose the pulp chamber. Following removal of the coronal pulp and achievement of homeostasis, a cotton pellet moistened with formocresol (1: 5 Buckley's solution) is placed on the amputated pulp for 5 min. The pulp stumps is then covered by IRM. After PP or FP treatment, all teeth are restored with a stainless steel crown.
* Follow-up: the follow-up for clinical and radiographic evaluation will be carried out at 6-month intervals. Treatment is considered a clinical failure if one or more of the following signs are observed: pain, abscess or sinus opening, tenderness upon percussion, or abnormal tooth mobility. For radiographic evaluation, the treatment is rated as a failure when one or more of the following signs are present: furcation or periapical radiolucency, pathologic external root resorption, or internal resorption. The treatment is regarded successful if both the clinical and radiographic evaluation does not indicate any signs of failure.

ELIGIBILITY:
Inclusion Criteria:

* The clinical criteria: primary molar with a deep carious lesion
* Sufficient tooth structure for restoration with a stainless steel crown
* No history of spontaneous pain
* Tenderness to percussion or abnormal mobility
* Abscess, fistula, or swelling of the gingiva, and with cessation of bleeding after a 2 mm depth of the pulp at the area of the exposure was amputated.
* The radiographic criteria: a deep carious lesion in close proximity to the pulp without furcation or radicular pathology
* Obliteration of the pulp and root canal, or internal or external root resorption.
* Physiologic root resorption, while included in the criteria, could not be more than one-third of the root length.

Exclusion Criteria:

* The clinical criteria: history of spontaneous pain
* Tenderness to percussion or abnormal mobility
* Abscess, fistula, or swelling of the gingiva, no cessation of bleeding after a 2 mm depth of the pulp at the area of the exposure was amputated.
* The radiographic criteria: tooth with furcation or radicular pathology
* Obliteration of the pulp and root canal, or internal or external root resorption.
* Physiologic root resorption more than one-third of the root length.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
partial pulpotomy clinical success rate | 6-month intervals, up to 2 years. From date of randomization until the date of first documented failure or up to 24 months
  Treatment is considered a clinical failure if one or more of the following signs are observed: pain, abscess or sinus opening, tenderness upon percussion, or abnormal tooth mobility. The treatment is regarded successful if clinical evaluation does not indicate any signs of failure.
partial pulpotomy radiographic success rate | 6-month intervals, up to 2 years. From date of randomization until the date of first documented failure or up to 24 months
  For radiographic evaluation, the treatment is rated as a failure when one or more of the following signs are present: furcation or periapical radiolucency, pathologic external root resorption, or internal resorption. The treatment is regarded successful if radiographic evaluation does not indicate any signs of failure.

SECONDARY OUTCOMES:
Formocresol pulpotomy clinical success rate | 6-month intervals, up to 2 years. From date of randomization until the date of first documented failure or up to 24 months
  Treatment is considered a clinical failure if one or more of the following signs are observed: pain, abscess or sinus opening, tenderness upon percussion, or abnormal tooth mobility. The treatment is regarded successful if clinical evaluation does not indicate any signs of failure.
Formocresol pulpotomy radiographic success rate | 6-month intervals, up to 2 years. From date of randomization until the date of first documented failure or up to 24 months
  For radiographic evaluation, the treatment is rated as a failure when one or more of the following signs are present: furcation or periapical radiolucency, pathologic external root resorption, or internal resorption. The treatment is regarded successful if radiographic evaluation does not indicate any signs of failure.